CLINICAL TRIAL: NCT01032421
Title: Gonadal Steroid Manipulation and Personality Characteristics: Association With Mood Fluctuations & IVF Outcomes
Brief Title: Gonadal Steroid Manipulation and Personality Characteristics: Association With Mood Fluctuations and in Vitro Fertilization (IVF) Outcomes
Acronym: IVF
Status: Completed | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Dr. Michal Roll, tel aviv souraski medical center
Other Study IDs: 04-284
Record Dates: First submitted 2009-11-25; First posted 2009-12-15 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Mood Disorders
Keywords: women admitted to the In Vitro Fertilization unit
MeSH Terms: conditions — Mood Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GNRH: Observational (IVF is not done as part of the study)
  Interventions: Procedure: IVF procedure

INTERVENTIONS:
Procedure: IVF procedure

SUMMARY:
The current study's primary aim is to investigate the association between neuroendocrine fluctuations and mood disorders by monitoring mood states over distinct hormonal phases during in-vitro-fertilization (IVF) treatment. The secondary goal of this study is to explore psychological profiles and coping mechanisms of women undergoing IVF, and to identify the ones that are associated with successful psychological adaptation to the process and a successful biological outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted for their first or second IVF cycle;
2. Demonstrated sufficient communication skills and level of understanding in the Hebrew language;
3. signed an informed consent;
4. Were under the age of 42;
5. Were not suffering from endometriosis or male factor in patients who underwent testicular sperm extraction (TESE);
6. Were not under psychotherapeutic or psychopharmacological treatment. The accepted indications for the IVF included a female factor, male factor or unexplained infertility.

Exclusion Criteria:

1. All others.

Max Age: 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women admitted for their first or second IVF cycle, under the age of 42. Please see the detailed inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

REFERENCES:
- [Derived] Zaig I, Azem F, Schreiber S, Amit A, Litvin YG, Bloch M. Psychological response and cortisol reactivity to in vitro fertilization treatment in women with a lifetime anxiety or unipolar mood disorder diagnosis. J Clin Psychiatry. 2013 Apr;74(4):386-92. doi: 10.4088/JCP.12m07805. PMID 23656846
- [Derived] Bloch M, Azem F, Aharonov I, Ben Avi I, Yagil Y, Schreiber S, Amit A, Weizman A. GnRH-agonist induced depressive and anxiety symptoms during in vitro fertilization-embryo transfer cycles. Fertil Steril. 2011 Jan;95(1):307-9. doi: 10.1016/j.fertnstert.2010.07.1073. PMID 20801439